CLINICAL TRIAL: NCT03559023
Title: A Factorial Trial of Ultrasound and Manometry to Improve the Success of Thoracic Epidural Placement
Acronym: USA-MAN-TE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Ivie, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18404
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Surgery
Keywords: Thoracic epidural
MeSH Terms: interventions — High-Energy Shock Waves; Manometry

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ultrasound Only (Active Comparator): Ultrasound assisted epidural placement
  Interventions: Procedure: Ultrasound Only
- Manometry Only (Active Comparator): Manometry confirmation in epidural placement
  Interventions: Procedure: Manometry Only
- Ultrasound Plus Manometry (Active Comparator): Ultrasound Plus Manometry confirmation in epidural placement
  Interventions: Procedure: Ultrasound Plus Manometry
- Usual Care/Management (Sham Comparator): Usual epidural technique placement
  Interventions: Procedure: Usual Care/Management

INTERVENTIONS:
Procedure: Ultrasound Only — The anesthesia team will use ultrasound to scan on subject's upper back (thoracic spine) to identify a place to begin the epidural procedure. A pen will be used to place markings on subject's back.
  Arms: Ultrasound Only
Procedure: Manometry Only — The anesthesia team will use an extra piece of tubing to confirm the epidural space one the epidural space is established.
  Arms: Manometry Only
Procedure: Ultrasound Plus Manometry — The anesthesia team will use both ultrasound and manometry to assist with epidural placement.
  Arms: Ultrasound Plus Manometry
Procedure: Usual Care/Management — The epidural will be placed using the usual technique utilized by the anesthesiology department. The the usual care/management group will receive a sham ("fake") ultrasound exam of subject's upper back with fake pen markings placed on subject's back. The ultrasound machine will not be turned on.
  Arms: Usual Care/Management

SUMMARY:
To investigate the use of ultrasound and manometry to increase the success rate of thoracic epidural placement. The use of ultrasound for lumbar epidural catheter placement is well established and is thought to assist in identifying an optimal skin entry point, depth to lamina and ligamentum flavum, and needle trajectory. The use of sterile manometry tubing to demonstrate a falling and oscillating fluid column has been described as a confirmatory test in the placement of lumbar epidurals. This study will determine if the efficacy of thoracic epidural placement is improved if placement is performed with the use of either US, or manometry, or both techniques combined, compared with a standard landmark-based placement technique alone.

DETAILED DESCRIPTION:
In a variety of thoracic and abdominal surgeries, thoracic epidural placement is associated with better pain relief, less opioid consumption, a decrease in adverse perioperative cardiac events, and improved intestinal perfusion and motility. Unfortunately, epidural catheter placement is challenging and is not always successful. The epidural space in the thoracic region is especially difficult to access due to the steep and inferior angulation of most of the spinous processes.

The vast majority of thoracic epidurals are placed using a landmark-based technique (i.e. without ultrasound guidance or fluoroscopy). In addition, a "loss of resistance" technique is typically used to confirm the needle has entered the epidural space. With a paramedian technique, the thoracic spinous processes are palpated (if possible), the needle is advanced through the skin just lateral to the spinous processes until lamina is contacted. The needle is then redirected medially based on an estimate of the location of the midline at the interlaminar space. The needle is then "walked" cephalad or caudad to blindly search for the interlaminar space. The depth to the lamina and interlaminar space are not known which introduces additional uncertainty in the mind of the operator, who must proceed with caution so as to not advance the needle too far and puncture the dural sac. It is not surprising that the landmark approach is associated with a significant number of unsuccessful attempts, long procedure times, and ineffective catheters, with the percentage of failed thoracic epidurals reported as high as 32%. In one study, the failure rate confirmed by both epidural waveform analysis and a sensory test after local anesthetic injection, the primary failure rate was found to be 23%-24%. A higher number of procedural attempts can also lead to an increased risk for complications including paresthesia, epidural hematoma, and dural puncture headaches. The high failure rate of this procedure highlights the need for more studies on ways to improve the techniques for thoracic epidural access.

Ultrasound (US) has proven to be useful in the imaging of the spine, and has also helped improve our ability to access the lumbar epidural space. Ultrasound measurement of the epidural space depth before epidural catheter placement decreased the rate of lumbar epidural catheter replacements, and reduced the number of epidural attempts when performed by first year residents compared to attempts without ultrasound guidance. In another study the use of ultrasound to identify the depth and location of the interlaminar and epidural space improved placement of labor epidurals with a lower number of block failures, a higher number of complete blockade, a higher rate of subject satisfaction, and lower VAS scores. Ultrasound has also been used to image the thoracic spine and epidural space.

The superior medial border of the thoracic transverse process aligns with the interlaminar space. This anatomical fact, combined with the ability to use ultrasound to identify the thoracic transverse processes and other bony landmarks forms the basis of this study. In the transverse plane, ultrasound can be used to identify the thoracic spinous processes and the midline. In the paramedian plane, the lamina, articular process and transverse process can be identified. In the lumbar spine, once the articular process is identified, a paramedian angulation of the ultrasound beam is used to identify an "acoustic window" between the lamina and into the spinal canal, thus identifying the interlaminar space. In the thoracic spine, because of the tight space between the lamina and overlapping of the lamina, an acoustic window is infrequently visualized and cannot be used as a reliable method to identify the interlaminar space. In contrast, both the superior border of the transverse process and the step-off between lamina can be readily identified with ultrasound. Both of these landmarks align with the interlaminar space.

In clinical practice, there is significant variability in techniques used to identify the correct epidural space. Although the loss of resistance technique is the most commonly used, variability exists in methods to confirm presence in the epidural space. Once such technique routinely used at this institution is the manometry technique. This involves using a three-way stopcock connected to clear plastic tubing IV extension tubing filled with normal saline. When the loss of resistance is detected, it can be confirmed by connecting the prefilled tubing to the Tuohy needle and opening the stopcock so the fluid inside is freely flowing. If the Tuohy needle tip is located in the epidural space, the saline column will initially fall, then exhibit pulsatility associated with heartbeat and respiration.

The identification of the epidural space by respiratory and heartbeat fluctuations in the air-fluid level has been previous described. The heart rate variability is believed to be due to arteriolar pulsations transmitted within a closed epidural space, while the respiratory variation in air fluid level is believed to be due to venous engorgement of the epidural veins with changes in thoracic pressure during inspiration. In the past 30 years, a handful of studies have been published evaluating epidural pressure measurement. Many of the studies using gravity to confirm presence in epidural space also use a pressure transducer to produce a visual waveform showing increase in pressure upon entry into the ligamentum flavum, and decrease in pressure upon entry into the epidural space. Two of these studies also incorporated an audible alarm to indicate change in pressure. One study correlated epidurals placed with pressure transducers to confirm the epidural space with presence or absence of block post-op and contrast spread on CT cathetergram showing a complete correlation between pressure waveform and catheter positioned in epidural space, further establishing the validity of pressure measurement to confirm entrance in the epidural space. Epidural pressure waveform analysis has not become routine practice, likely due to equipment, cost, and time constraints. We hypothesize that the simple, rapid, and inexpensive technique of extension tubing manometry will offer similar benefits for confirmation of epidural placement and will be applicable to placement at the thoracic levels.

ELIGIBILITY:
Inclusion Criteria:

* Epidural indicated for a T4-T10 placement site
* American Society of Anesthesiologists (ASA) physical status I to IV

Exclusion Criteria:

* Non-English speaking subjects in situations when an interpreter or consent in their native language is not available.
* Pregnant women
* Decsionally impaired
* Prisoners
* Children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Successful thoracic epidural placement | 15 minutes after injection of 1.5% lidocaine
  Successful thoracic epidural placement as measured by diminished sensation to pinprick in two or more adjacent dermatomes 15 minutes after the injection of 5 mL of 1.5% lidocaine with 1:200,000 epinephrine into an epidural catheter.

SECONDARY OUTCOMES:
Diminished sensation to cold | 15 minutes after injection of lidocaine
  Diminished sensation to cold in two or more adjacent dermatomes 15 minutes after the injection of 5 mL of 1.5% lidocaine with 1:200,000 epinephrine into an epidural catheter.
Average pain score | First 24 hours postoperatively
  Mean pain scores documented in the electronic medical record
Number of attempts | During epidural placement
  Number of times the Tuohy needle is withdrawn to skin and re-inserted
Procedure time | During epidural placement
  Time from start of local anesthetic infiltration to the time of Tuohy withdrawal
Complications | During epidural placement
  Dural puncture, positive test response

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Ivie, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States